CLINICAL TRIAL: NCT05442281
Title: Vegan Diet in Young Children - Studies of Nutritional Intake, Growth and Neurodevelopment
Brief Title: Vegan Diet in Small Children
Acronym: VHS
Status: Recruiting | Type: Observational
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Staffan Berglund, Senior Consultant, associate professor, Umeå University
Other Study IDs: VHS
Record Dates: First submitted 2022-05-23; First posted 2022-07-01 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Vegan Diet

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, breast milk, whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Vegan diet: Children fed vegan diet from 6 months of life
- Mixed diet: Children fed mixed diet from 6 months of life

SUMMARY:
Following increased knowledge about climate change and how food production affects greenhouse gas emissions, the interest in vegetarian diets is increasing. In line with this, also vegan diet is becoming more common at all ages, including in young children. But the state of knowledge regarding the effect of this diet on children during infancy and early childhood has been poorly studied and existing literature consists to a large extent of case reports.

With the main hypothesis that vegan diet from the introduction of complementary foods causes reduced bio availability of certain micronutrients important for development, the aim of this study is to examine dietary intake and development during the first years of life in a group of children eating vegan diet and compare with a reference group eating mixed diets.

In an observational study, investigators plan to include 30 children before the age of 6 months during the years 2021-2026, where the parents have decided to offer their child only vegan food. The children are studied in comparison with a reference group of 30 matched cases regarding growth, nutritional status, and dietary intake. Data collection includes monthly dietary records and blood sample analyses and growth at 6, 12 and 24 months. At the age of 3, cognitive developmental assessment (WPSSI-IV) and an DEXA examination of body composition are performed.

The study is expected to contribute to increased knowledge about the risk and benefits of vegan diets and thereby provide a better basis for future recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Planned exclusive vegan diet or mixed diet respectively from 6 months of age until at least 2 years of life
* Exclusively (>90%) breastfed until 4 months
* Born term (GE 37+0 - 41+6)
* Single birth
* Birth weight >2500 g
* Apgar score 5 min > 5

Exclusion Criteria:

* A chronic disease affecting growth or neurodevelopment

Ages: 4 Months to 8 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Swedish infants mainly breastfed planned for vegan or mixed diet respectively
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Concentration of Hemoglobin | 12 months of age
  Blood
Body Weight (kg) | 12 months of age
  measured weight at 12 mo using a device for measuring weight

SECONDARY OUTCOMES:
Wechsler Preschool & Primary Scale of Intelligence | 3 years of age
  Scale for cognitive development. Expected mean 100. Higher scores equals better cognitive development.
Fat mass index | 3 years of age
  FMI, measured by DEXA-scan
Lean mass index | 3 years of age
  LMI, measured by DEXA-scan
Protein intake | at 12 months of age
  3 day food diary
Fat intake | at 12 months of age
  3 day food diary
Carbohydrate intake | at 12 months of age
  3 day food diary
Iron intake (mg/day) | throughout study
  3 day food diary
B12 levels | 6, 12, 24, 36 months
  Serum sample
Zink level | 6, 12, 24, 36 months
  Serum sample
D-vitamin levels | 6, 12, 24, 36 months
  Serum sample
Calcium levels | 6, 12, 24, 36 months
  Serum sample
Homocysteine levels | 6, 12, 24, 36 months
  serum sample
Transferrin receptor concentration | 12 months of age
  Serum sample
Transferrin saturation | 12 months of age
  serum sample
Mean cell volume | 12 months of age
  Blood sample
Ferritin | 12 months of age
  Serum sample
Length of body | 12 months of age
  measured length at 12 mo using measuring tool for children
Circumference of the head | 12 months of age
  measured at 12 mo using measuring tool for children

CONTACTS AND LOCATIONS:
Locations (1):
- Umeå University, Department of Clinical Sciences, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: No